CLINICAL TRIAL: NCT02382107
Title: A Blinded, Cross-sectional, Diagnostic Evaluation Study Performed in Pulmonary TB Suspects at the TB Dispensary for Sector 4 of the Marius-Nasta-Institute in Bucharest, Romania
Status: Completed | Type: Observational
Sponsor: Michael Hoelscher (Other)
Collaborators: "Marius Nasta" Pulmonology Institute (Other); Clinical Infectious Diseases Research Center Borstel, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Chief Investigator, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-Bucharest-01
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Tuberculosis
Keywords: TB; Tuberculosis; Diagnostic study
MeSH Terms: conditions — Tuberculosis; Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, urine, sputum
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational — TB suspects, who present themselves to the pulmonary ambulance at the Marius Nasta Instiute

SUMMARY:
The diagnosis of tuberculosis (TB) and especially the detection of drug resistance of tuberculosis mycobacteria can be time consuming and costly. New and rapid diagnostic tests are needed to improve early case detection and correct initiation of treatment.

In the planned cross-sectional diagnostic evaluation study the investigators are aiming for the assessment of several new TB diagnostics (e.g. new AID strip assays and TrDNA assay in urine) in TB suspects who are presenting themselves to the pulmonary ambulance (TB dispensary for sector 4) at the Marius Nasta Institute (MNI). The study will be conducted in a co-operation between the MNI and the German Center for Infection Research (DZIF).

DETAILED DESCRIPTION:
Up to 400 TB suspects will be consecutively screened for their eligibility for participation in the study. In those who are eligible (according to the criteria listed above) to participate, 2 sputum samples and one urine will be collected for standard diagnostic testing for TB in sputum (smear, Line Probe Assays and culture methods, as defined in the national guidelines) and for the evaluation of the new assays; one blood sample will be collected for analysis of lipoprotein profiles in serum of TB patients. Further, a HIV test and a clinical examination will be performed in all study subjects. Information on risk factors for TB disease (co-morbidities such as diabetes mellitus, co-medication such as steroids and risk behaviour such as smoking) will be also documented.

All TB tests results and data which are generated in the study will be collected on standardized study forms and entered in a password-secured data base. TB tests results will be also shared with the medical staff treating the patients who are participating in the study.

One follow up visit will be performed after 8 weeks in order to evaluate the clinical progress of the participants, either on TB treatment (if TB was confirmed) or alternative therapy, in participants who were not diagnosed with TB.

The isolated TB strains will be sent to the Research Center Borstel in Germany for evaluation through sequencing and phenotypic methods. The remnants of collected samples will be stored in the National TB Laboratory for future evaluations of new tests.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected pulmonary TB, who have a chest radiograph which is compatible with pulmonary TB plus one of the signs or symptoms listed below and indicative of possible TB:
* Productive cough for more than 2 weeks
* Haemoptysis
* Fever
* Night sweats
* Substantial involuntary weight loss
* Subject able and willing to give informed consent, including for HIV-testing

Exclusion Criteria:

* anti-tuberculosis therapy with simultaneous administration of at least 2 active compounds taken currently or within the previous 6 months
* physical or mental inability preventing study participation as determined at the discretion of the investigator
* member of a vulnerable population group (prisoner, soldier, mental illness, under guardianship, age <18 years)
* extrapulmonary tuberculosis without pulmonary involvement
* incapability to produce 2 sputum samples of sufficient quality (mucoid) and volume (at least 3ml)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TB suspects who presented themselves to the pumonology ambulatory at the Marius Nasta Institute
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The main objective is the evaluation of the diagnostic characteristics (sensitivity, specificity) of several new rapid diagnostic tests for TB compared to culture (both liquid and solid) as the reference standard in patients | Up to 70 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Elmira Ibraim, MD, Principal Investigator — Marius Nasta Pulmonology Institute, Sos. Viilor 90 Sector 5, 050159 Bucharest, Romania
Locations (1):
- Marius Nasta Pulmonology Institute, Bucharest, Romania